CLINICAL TRIAL: NCT05603156
Title: A Prospective, Single-arm, Multi-center Study of Olverembatinib Combined With Inotuzumab Ozogamicin in the Treatment ph+ ALL With MRD Persistent Positive
Brief Title: A Study of Olverembatinib Combined With Inotuzumab Ozogamicin in the Treatment ph+ ALL With MRD Persistent Positive
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022033
Record Dates: First submitted 2022-10-24; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Ph+ ALL; Bone Marrow Transplant; Minimal Residual Disease
Keywords: ph+ALL; HSCT; MRD persistent positive; Inotuzumab; tyrosine kinase inhibitor
MeSH Terms: conditions — Neoplasm, Residual | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): patients enrolled treated with the combination of Olverembatinib and Inotuzumab to clear the persistent MRD.
  Interventions: Drug: the usage of Olverembatinib combined with Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: the usage of Olverembatinib combined with Inotuzumab Ozogamicin — patients in this arm will accept a 28 days treatment regimen: Olverembatinib 40mg QOD (d1 to d28 )and Inotuzumab Ozogamicin 1.2mg/m2 (divided into 2 days, d1 and d8, 0.6mg/m2, respectively).

SUMMARY:
Hematopoietic stem cell transplantation (HSCT) is the effective and even the only cure treatment option for ph+ acute lymphocyte leukemia (ph+ALL). However, the outcome has been insufficient and relapse remains the major cause of treatment failure and poor survival, especially for patients with persistent minimal residual disease (MRD). It is believed that clearance of MRD pre-HSCT could significantly reduce the incidence of relapse post-HSCT. Olverembatinib has been documented as a promising third generation of TKIs. Meanwhile, Inotuzumab ozogamicin (InO) , an antibody-drug conjugate approved in the US and the European Union, has been applied in relapsed/refractory acute lymphoblastic leukemia (R/R ALL) and achieved good treatment outcome. This prospective, single arm and multicenter study is to investigate the efficacy and safety of combination of Olverembatinib and Ino for MRD clearance before bridging to HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Acute lymphoblastic leukemia with positive Ph chromosome or BCR / ABL fusion gene ; cD22 expression on the surface of leukemia cells ; hematological complete remission but with MRD persistent positive ( BCR-ABL1 level ≥ 10-4 ), after at least 3 times of intensive chemotherapy, in which classical chemotherapy combined with any first or second generation of tyrosine kinase inhibitors targeting BCR-ABL1.
2. Be ≥ 18 years of age on the day of enrollment.
3. Understand the study procedures, alternative treatment available, and risks involved with the study, and voluntarily agree to participate by giving written informed consent.
4. Necessary to meet the criteria of important organ function : renal function and liver function are as follows : AST, ALT and ALP below the normal 2 times the upper limit, total bilirubin below the normal upper limit 1.5 times ; creatinine clearance rate greater than 50ML / min ; pancreatic function : serum amylase is not higher than the normal upper limit 1.5 times, serum lipase is not higher than the normal upper limit 1.5 times ; normal heart function : ejection fraction ( EF ) > 60 %, pulmonary artery systolic pressure ≤ 50mmHg.
5. Has documented nefative results for human immunodeficiency virus antibody (HIV-Ab), hepatitis C virus antibody (HCV-Ab) , as well as undetectable HCV RNA, or undetectable HBV DNA.
6. ECOG-PS 0-2.
7. Informed consent must be signed before the start of the trial. Informed consent must be signed by the patient himself or his direct family members who are 18 years old and above ; considering the patient 's condition, if the patient 's signature is not conducive to the treatment of the disease, the informed consent is signed by the legal guardian or the patient 's immediate family.

Exclusion Criteria:

1. Diagnosed as mixed lineage leukemia.
2. Documented as CNS leukemia or extramedullary infiltration.
3. Patients with other malignant tumors ; the patients were assessed as having comorbidities that seriously endanger the patient 's life or affect the patient 's completion of the study.
4. Used to use the third generation of TKIs, including Olverembatinib.
5. Patients received any other kind of anti-leukemia antibody therapy two weeks before enrollment.
6. Patients received radiotherapy or chemotherapy (except induction chemotherapy ) or any other research treatment within two weeks before enrollment, with the following exceptions :Designed to reduce circulating leukemia lymphocytes count or remission : Steroids, hydroxyurea or vincristine;Maintenance therapy : thiopurine, methotrexate, vincristine, thioguanine and / or tyrosine kinase inhibitors.
7. Patients with severe allergies to InO components and excipients ( Grade ≥ 3 ).
8. History of clinically significant liver disease, such as hepatic veno - occlusive disease ( VOD ) or sinusoidal obstruction syndrome ( SOS ) ; such as cirrhosis, decompensated liver disease, acute or chronic hepatitis.
9. Active heart disease, defined as one or more of the following : with any history of heart or vascular disease ; have uncontrolled or symptomatic angina history ; myocardial infarction less than 6 months before enrollment ; a history of arrhythmia requiring drug treatment or severe clinical symptoms ; uncontrolled or symptomatic congestive heart failure ( > NYHA grade 2 ) ; ejection fraction is below the lower limit of the normal range. Cardiac ultrasound pulmonary artery systolic pressure > 50mmHg ; or pulmonary hypertension - related clinical symptoms.
10. Severe cardiovascular disease, including myocardial infarction, unstable angina, severe arrhythmia, congestive heart failure, etc. during previous TKI treatment.
11. A history of auto- or allo-HSCT.
12. Dysfunction of blood coagulation.
13. Positive serological response to known HIV or active hepatitis C virus.
14. Patients with mental illness or other conditions that do not meet the requirements of research treatment and monitoring.
15. Unable or unwilling to sign consent form.
16. Pregnant or lactating women.
17. Patients with other special conditions assessed as unqualified by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
MRD clearance rate | 2 weeks after the treatment with Olverembatinib and Inotuzumab Ozogamicin
  The ratio of patients achieved MRD remission. The MRD remission was defined as the fusion gene BCR-ABL quantification in bone marrow samples was lower than the detection limit of RT-PCR ( < 0.01 %, the residual number of leukemia cells detected in our hospital was 0.0032 % ) ; at the same time, flow cytometry ( FACS ) was used to monitor the MRD of the cells, and the proportion of abnormal cells < 0.1 % was MRD-

SECONDARY OUTCOMES:
One year OS after HSCT | One year after HSCT
  For patients achived MRD remission, HSCT will be performed. The one year overall survival after HSCT will be the seconday outcom.
One year RFS after HSCT | One year after HSCT
  For patients achived MRD remission, HSCT will be performed. The one year relaspe free survival after HSCT will be the seconday outcom.
One year NRM after HSCT | One year after HSCT
  For patients achived MRD remission, HSCT will be performed. The one year non-relaspe mortality after HSCT will be the seconday outcom.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No